CLINICAL TRIAL: NCT01838031
Title: Randomized Thyroid Screening Protocol During Pregnancy: a Multi-center Prospective Controlled Study
Brief Title: Thyroid Screening Protocol During Pregnancy: a Multi-center Prospective Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Liangkun Ma, associate profesoor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Z111107058811025
Record Dates: First submitted 2013-04-14; First posted 2013-04-23 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Subclinical Hypothyroidism
Keywords: antenatal thyroid screening; subclinical hypothyroidism; thyroid function; thyroid antibody; pregnancy outcome; childhood cognitive function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the control group (No Intervention): The serum will be stored and the measurements will be obtained after the delivery
- the thyroid screening group (Active Comparator): The thyroid function and antibody will be measured during pregnancy. The subclinical hypothyroidism will be treated individually.
  Interventions: Other: thyroid screening

INTERVENTIONS:
Other: thyroid screening — The thyroid function and antibody will be measured immediately. The subclinical hypothyroidism will be treated individually.
  Arms: the thyroid screening group

SUMMARY:
Estimate the proper thyroid screening method during pregnancy. Evaluate if maternal subclinical hypothyroidism treatment during pregnancy result in improved pregnancy outcome and cognitive function in the children.

DETAILED DESCRIPTION:
The investigators conducted a single-blinded trial in which pregnant women at a gestation of less than 12 weeks, usually 6 to 8 weeks, provided blood samples for measurement of thyrotropin, free thyroxine(FT4) and thyroid peroxidase antibody (TPOAb). Women were assigned to a screening group in PUMCH (in which measurements were obtained immediately) or a control group in HMCHH (in which serum was stored and measurements were obtained shortly after delivery). Each group enrolled 1000 pregnant women separately. Women with positive findings in the screening group were given individualized levothyroxine treatment and regular follow-up. Compare the pregnancy outcomes, IQ at 2-3 years of age in children of women with subclinical hypothyroidism between two groups.

ELIGIBILITY:
Inclusion Criteria:

* All of the pregnant women who receive prenatal care in PUMCH and HMCHH
* Sign the consent form
* agree to follow-up the pregnancy outcome and child

Exclusion Criteria:

* the pregnant women who do not agree to enter the study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 1 year
  the number of miscarriage，preeclampsia，gestational diabetes，prererm birth and postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Bahn Chair RS, Burch HB, Cooper DS, Garber JR, Greenlee MC, Klein I, Laurberg P, McDougall IR, Montori VM, Rivkees SA, Ross DS, Sosa JA, Stan MN; American Thyroid Association; American Association of Clinical Endocrinologists. Hyperthyroidism and other causes of thyrotoxicosis: management guidelines of the American Thyroid Association and American Association of Clinical Endocrinologists. Thyroid. 2011 Jun;21(6):593-646. doi: 10.1089/thy.2010.0417. Epub 2011 Apr 21. PMID 21510801
- [Background] Lazarus JH, Bestwick JP, Channon S, Paradice R, Maina A, Rees R, Chiusano E, John R, Guaraldo V, George LM, Perona M, Dall'Amico D, Parkes AB, Joomun M, Wald NJ. Antenatal thyroid screening and childhood cognitive function. N Engl J Med. 2012 Feb 9;366(6):493-501. doi: 10.1056/NEJMoa1106104. PMID 22316443